CLINICAL TRIAL: NCT01505257
Title: Early Nurse Detection of Delirium Superimposed on Dementia
Brief Title: Early Nurse Detection and Management of Delirium
Acronym: END-DSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Vanderbilt University Medical Center (Other); Harvard University (Other); Augusta University (Other)
Responsible Party: Principal Investigator, Donna Fick, PhD, RN, FGSA, FAAN, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01NR011042 (NIH)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Delirium Superimposed on Dementia
Keywords: Delirium; Dementia; Confusion Assessment Method
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- END-DSD Intervention (Experimental)
  Interventions: Behavioral: END-DSD
- Control (No Intervention)

INTERVENTIONS:
Behavioral: END-DSD — Multi-component intervention including 1) Nursing education regarding detection and management of delirium superimposed on dementia; 2) Computerized decision support and EHR; 3) A unit champion nurse for promotion of delirium assessment and management; 4) Feedback to nursing staff
  Arms: END-DSD Intervention

SUMMARY:
Delirium (acute confusion) is common and costly in persons with dementia, resulting in longer hospital stays, more complications, and greater functional decline. This research tests the use of the electronic health record, education, and regular feedback to nurses to improve detection and management of delirium. Ultimately, findings will direct ways to improve acute care of this vulnerable population.

DETAILED DESCRIPTION:
Delirium is an acute, reversible change in mental status that occurs in over 40% of persons with dementia. Delirium superimposed on dementia (DSD) leads to increased mortality, increased costs, nursing home placement, early re-hospitalization, and functional decline. Delirium in persons with dementia appears to substantially worsen outcomes in persons with dementia- who are already burdened with functional decline. The purpose of this study is to improve nursing detection and management of delirium in persons with dementia and decrease the duration and patient complications of delirium. To achieve these objectives, a multi-component intervention strategy called, Early Nurse Detection of Delirium Superimposed on Dementia (END DSD) will be tested. END-DSD employs a paired cluster randomized trial (C-RCT) of three hospitals with a total of six inpatient units and 360 hospitalized persons with dementia to achieve these objectives. END DSD intervention consists of 1) Nursing education regarding DSD, 2) Computerized decision support through standardized delirium assessment and management screens via the electronic health record (EHR), 3) an identified unit champion on each intervention unit who will be utilized to persuade other nurses to implement the innovation, and 4) Weekly feedback to the nursing staff to further facilitate assessment and management of delirium. We are testing the following specific aims: A.1: To determine whether the intervention "END DSD" improves nurse detection and management of DSD. A.2: To determine the effect of "END DSD" intervention on patient clinical outcomes, including duration of delirium and rate of psychoactive medications.

The study focuses on a costly and prevalent problem, and utilizes a novel approach that via the EHR will clearly be replicable across settings of care. END-DSD has the potential to significantly improve quality of life and decrease costs of care by: improving the detection of DSD; increasing the use of non-pharmacological management of DSD; shortening the duration of delirium and hospital length of stay; and decreasing the use of inappropriate medications, thus mitigating the complications of DSD. This project builds on over a decade of funded research and clinical practice by the investigators, and brings their unique and collaborative efforts together in an innovative manner to impact the under addressed problem of DSD in hospitalized older adults.

ELIGIBILITY:
Inclusion Criteria:

* Persons with dementia will be included if they: a) are on one of the selected medical-surgical units and are age 65 years or older; b) have been hospitalized less than 48 hours; and c) meet the criteria for dementia. The study will include minorities and women.

Exclusion Criteria:

* Persons with dementia will be excluded if they have any significant neurological or neurosurgical disease associated with cognitive impairment other than dementia (due to confounding with dementia or DSD), such as:

  * Lewy Body Dementia
  * Huntington's disease
  * Sormal pressure hydrocephalus
  * Seizure disorder
  * Subdural hematoma
  * Head trauma
  * Known structural brain abnormalities
* Nonverbal and unable to communicate due to severe dementia (MMSE=0)
* Aphasia
* Intubation
* Terminal illness (since interviews are required for the study).
* This study will not exclude persons with pre-existing delirium.
* In addition, subjects will not be excluded on the basis of race or gender.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 391 (Actual)
Dates: Start 2010-04; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Severity of Delirium | Participants will be assessed daily until discharge (duration of hospitalization), which is expected to be about 5 days
  Measured using the Delirium Rating Scale R-98.
Inappropriate CNS-Active Medication Use | Participants will be assessed daily until discharge (duration of hospitalization), which is expected to be about 5 days
  Ascertained from patient's medical record
Nurse Detection of Delirium | Participants will be assessed every shift until discharge (duration of hospitalization), which is expected to be about 5 days
  Ascertained through electronic health record and chart review
Delirium Duration | Participants will be assessed daily until discharge (duration of hospitalization), which is expected to be about 5 days
  Measured using the Confusion Assessment Method (CAM)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Fick, RN,PhD, Principal Investigator — Penn State University; Lorraine Mion, RN,PhD, Study Chair — Vanderbilt University; Jane McDowell, MSN, Study Director — Penn State University; Sharon Inouye, MD, MPH, Study Chair — Harvard University; Ann Kolanowski, RN,PhD,FAAN, Study Chair — Penn State University
Locations (2):
- United States (2):
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee